CLINICAL TRIAL: NCT01716234
Title: Phase 1B Study of the Safety, Tolerance, and Pharmacokinetics of Oral Posaconazole in Immunocompromised Children With Neutropenia (P03579)
Brief Title: A Study of the Safety, Tolerance, and Pharmacokinetics of Oral Posaconazole in Immunocompromised Children (P03579)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was terminated early (10 July 2015) based on preliminary analysis of pharmacokinetic data.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P03579; 2007-004645-15 (EudraCT Number); MK-5592-032 (Other: Merck)
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Results first posted 2016-04-15 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Fungal Infections
MeSH Terms: conditions — Mycoses | interventions — posaconazole; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- POS 12 BID 2 to <7 Years (Experimental): Participants aged 2 to <7 years received posaconazole oral suspension 12 mg/kg/day divided into 2 doses (BID) until recovery from neutropenia or up to 28 days.
  Interventions: Drug: Posaconazole 12 mg/kg/day BID
- POS 12 BID 7 to <18 Years (Experimental): Participants aged 7 to <18 years received posaconazole oral suspension 12 mg/kg/day divided into 2 doses (BID) until recovery from neutropenia or up to 28 days.
  Interventions: Drug: Posaconazole 12 mg/kg/day BID
- POS 18 BID 2 to <7 Years (Experimental): Participants aged 2 to <7 years received posaconazole oral suspension 18 mg/kg/day divided into 2 doses (BID) until recovery from neutropenia or up to 28 days.
  Interventions: Drug: Posaconazole 18 mg/kg/day BID
- POS 18 BID 7 to <18 Years (Experimental): Participants aged 7 to <18 years received posaconazole oral suspension 18 mg/kg/day divided into 2 doses (BID) until recovery from neutropenia or up to 28 days.
  Interventions: Drug: Posaconazole 18 mg/kg/day BID
- POS 18 TID 2 to <7 Years (Experimental): Participants aged 2 to <7 years received posaconazole oral suspension 18 mg/kg/day divided into 3 doses (TID) until recovery from neutropenia or up to 28 days.
  Interventions: Drug: Posaconazole 18 mg/kg/day TID
- POS 18 TID 7 to <18 Years (Experimental): Participants aged 7 to <18 years received posaconazole oral suspension 18 mg/kg/day divided into 3 doses (TID) until recovery from neutropenia or up to 28 days.
  Interventions: Drug: Posaconazole 18 mg/kg/day TID
- POS 12 TID 3 months to <2 Years (Experimental): Participants aged 3 months to <2 years received posaconazole oral suspension 12 mg/kg/day divided into 3 doses (TID) until recovery from neutropenia or up to 28 days.
  Interventions: Drug: Posaconazole 12 mg/kg/day TID

INTERVENTIONS:
Drug: Posaconazole 12 mg/kg/day BID — Posaconazole oral suspension 12 mg/kg/day divided into 2 doses (BID) (maximum 800 mg/day)
  Other Names: SCH 056592; MK-5592; Noxafil®
  Arms: POS 12 BID 2 to <7 Years; POS 12 BID 7 to <18 Years
Drug: Posaconazole 18 mg/kg/day BID — Posaconazole oral suspension 18 mg/kg/day divided into 2 doses (BID) (maximum 1200 mg/day)
  Other Names: SCH 056592; MK-5592; Noxafil®
  Arms: POS 18 BID 2 to <7 Years; POS 18 BID 7 to <18 Years
Drug: Posaconazole 18 mg/kg/day TID — Posaconazole oral suspension 18 mg/kg/day divided into 3 doses (TID) (maximum 1200 mg/day)
  Other Names: SCH 056592; MK-5592; Noxafil®
  Arms: POS 18 TID 2 to <7 Years; POS 18 TID 7 to <18 Years
Drug: Posaconazole 12 mg/kg/day TID — Posaconazole oral suspension 12 mg/kg/day divided into 3 doses (TID) (maximum 800 mg/day)
  Other Names: SCH 056592; MK-5592; Noxafil®
  Arms: POS 12 TID 3 months to <2 Years

SUMMARY:
The purpose of this dose-escalation study is to evaluate the pharmacokinetics, safety, and tolerability of oral posaconazole in immunocompromised children with neutropenia or expected neutropenia.

ELIGIBILITY:
Inclusion Criteria:

* Documented or anticipated neutropenia expected to last at least 7 days and only in the following clinical situations: acute leukemia; myelodysplasia; severe aplastic anemia; autologous hematopoietic stem cell transplantation (HSCT) recipients; high risk neuroblastoma; advanced stage non-Hodgkin's lymphoma; recipients of allogeneic HSCT during the pre-engraftment (neutropenia) period
* Participants of child-bearing potential must use a medically accepted method of

contraception throughout the study and for at least 30 days after stopping study medication, unless they are surgically or medically sterile or agree to remain abstinent.

Exclusion Criteria:

* Proven invasive fungal infection (IFI) before study entry
* Severe nausea and/or vomiting at screening
* Received posaconazole within 10 days before screening
* Unable to receive study drug by mouth or via an intestinal (enteral) tube
* Females who are pregnant, intend to become pregnant during the study, or are breastfeeding
* History of anaphylaxis attributed to the azole class of antifungal agents

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 142 (Actual)
Dates: Start 2008-04-17 (Actual); Primary Completion 2015-04-01 (Actual); Study Completion 2015-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Arrieta AC, Sung L, Bradley JS, Zwaan CM, Gates D, Waskin H, Carmelitano P, Groll AH, Lehrnbecher T, Mangin E, Joshi A, Kartsonis NA, Walsh TJ, Paschke A. A non-randomized trial to assess the safety, tolerability, and pharmacokinetics of posaconazole oral suspension in immunocompromised children with neutropenia. PLoS One. 2019 Mar 26;14(3):e0212837. doi: 10.1371/journal.pone.0212837. eCollection 2019. PMID 30913226

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 160 participants were screened, 142 were randomized / enrolled, and 136 were treated. An arm planned for participants aged 3 months to <2 years to receive posaconazole 18 mg/kg/day TID was never initiated.
Period: Overall Study
Arm/Group | POS 12 BID 2 to <7 Years | POS 12 BID 7 to <18 Years | POS 18 BID 2 to <7 Years | POS 18 BID 7 to <18 Years | POS 18 TID 2 to <7 Years | POS 18 TID 7 to <18 Years | POS 12 TID 3 Months to <2 Years
Started | 24 | 22 | 20 | 28 | 15 | 32 | 1
Treated | 22 | 21 | 19 | 28 | 15 | 30 | 1
Completed | 14 | 12 | 15 | 16 | 10 | 18 | 1
Not Completed | 10 | 10 | 5 | 12 | 5 | 14 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 1 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Did not meet protocol eligibility | 0 | 0 | 1 | 0 | 0 | 4 | 0
Not completed — Adverse Event | 7 | 10 | 2 | 8 | 3 | 6 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 2 | 2 | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | POS 12 BID 2 to <7 Years | POS 12 BID 7 to <18 Years | POS 18 BID 2 to <7 Years | POS 18 BID 7 to <18 Years | POS 18 TID 2 to <7 Years | POS 18 TID 7 to <18 Years | POS 12 TID 3 Months to <2 Years | Total
Number analyzed (Participants) | 24 | 22 | 20 | 28 | 15 | 32 | 1 | 142
Age, Continuous [Mean (Standard Deviation); unit: Years] | 4.0 (1.3) [2 to 7] | 11.9 (3.5) [7 to 17] | 4.4 (1.5) [2 to 7] | 12.2 (3.2) [7 to 18] | 4.1 (1.3) [3 to 7] | 13.1 (3.0) [7 to 18] | 0.9 (0) [1 to 1] | 8.9 (4.9) [1 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 8 | 9 | 6 | 14 | 0 | 59
  Male | 14 | 10 | 12 | 19 | 9 | 18 | 1 | 83

OUTCOME MEASURES:

1. Primary Outcome: Average Concentration of Posaconazole (Cavg) on Day 1 (Single Dose)
Description: Blood samples for determination of plasma posaconazole concentration were collected predose and approximately 3, 5, 8, and 12 hours after the first dose on Day 1. The 12-hour sample was not obtained for the TID dose groups. Day 1 pharmacokinetic samples were not collected for participants 3 months to <2 years of age weighing <6.5 kg.
Time Frame: Up to 12 hours after the first dose (BID dose groups) or up to 8 hours after the first dose (TID dose (TID dose groups)
Population: The pharmacokinetic evaluable population included all treated participants with evaluable samples applicable to the endpoint.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | POS 12 BID 2 to <7 Years | POS 12 BID 7 to <18 Years | POS 18 BID 2 to <7 Years | POS 18 BID 7 to <18 Years | POS 18 TID 2 to <7 Years | POS 18 TID 7 to <18 Years | POS 12 TID 3 Months to <2 Years
Number analyzed (Participants) | 22 | 19 | 12 | 12 | 5 | 10 | 1
ng/mL | 122 (101) | 107 (92.5) | 112 (86.9) | 113 (100) | 68.4 (40.4) | 57.9 (30.2) | 68.5 (0)

2. Primary Outcome: Average Concentration of Posaconazole (Cavg) on Day 7 (Steady State)
Description: Blood samples for determination of plasma posaconazole concentration were collected predose and approximately 3, 5, 8, and 12 hours after the first dose on Day 7 (steady state). The 12-hour sample was not obtained for the TID dose groups. The target Cavg range was 500 to <2500 ng/mL.
Time Frame: Up to 12 hours after the first dose on Day 7 (BID dose groups) or up to 8 hours after the first dose on Day 7 (TID dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | POS 12 BID 2 to <7 Years | POS 12 BID 7 to <18 Years | POS 18 BID 2 to <7 Years | POS 18 BID 7 to <18 Years | POS 18 TID 2 to <7 Years | POS 18 TID 7 to <18 Years | POS 12 TID 3 Months to <2 Years
Number analyzed (Participants) | 16 | 14 | 12 | 12 | 5 | 10 | 1
ng/mL | 604 (779) | 1050 (789) | 485 (306) | 1240 (1400) | 620 (411) | 1150 (750) | 453 (0)

3. Secondary Outcome: Number of Participants With an Adverse Event
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product, biologic (at any dose), or medical device, which does not necessarily have a causal relationship with the treatment. Adverse events may include the onset of new illness and the exacerbation of preexisting conditions.
Time Frame: Up to Day 58
Population: The population analyzed was all treated participants.
Measure: Number; unit: Participants
Arm/Group | POS 12 BID 2 to <7 Years | POS 12 BID 7 to <18 Years | POS 18 BID 2 to <7 Years | POS 18 BID 7 to <18 Years | POS 18 TID 2 to <7 Years | POS 18 TID 7 to <18 Years | POS 12 TID 3 Months to <2 Years
Number analyzed (Participants) | 22 | 21 | 19 | 28 | 15 | 30 | 1
Participants | 21 | 21 | 16 | 26 | 13 | 30 | 1

4. Secondary Outcome: Number of Participants With an Adverse Event Leading to Study Drug Discontinuation
Description: as for outcome 3
Time Frame: Up to Day 28
Population: The population analyzed was all treated participants.
Measure: Number; unit: Participants
Arm/Group | POS 12 BID 2 to <7 Years | POS 12 BID 7 to <18 Years | POS 18 BID 2 to <7 Years | POS 18 BID 7 to <18 Years | POS 18 TID 2 to <7 Years | POS 18 TID 7 to <18 Years | POS 12 TID 3 Months to <2 Years
Number analyzed (Participants) | 22 | 21 | 19 | 28 | 15 | 30 | 1
Participants | 7 | 9 | 2 | 9 | 3 | 6 | 0

ADVERSE EVENTS:
Time Frame: All AEs: from Day 1 up to Day 39; SAEs: up to Day 58.
Description: The population analyzed is all treated participants.
Groups:
- POS 12 BID 2 to <7 Yrs: Participants aged 2 to <7 years received posaconazole oral suspension 12 mg/kg/day divided into 2 doses (BID) until recovery from neutropenia or up to 28 days.
- POS 12 BID 7 to <18 Yrs: Participants aged 7 to <18 years received posaconazole oral suspension 12 mg/kg/day divided into 2 doses (BID) until recovery from neutropenia or up to 28 days.
- POS 18 BID 2 to <7 Yrs: Participants aged 2 to <7 years received posaconazole oral suspension 18 mg/kg/day divided into 2 doses (BID) until recovery from neutropenia or up to 28 days.
- POS 18 BID 7 to <18 Yrs: Participants aged 7 to <18 years received posaconazole oral suspension 18 mg/kg/day divided into 2 doses (BID) until recovery from neutropenia or up to 28 days.
- POS 18 TID 2 to <7 Yrs: Participants aged 2 to <7 years received posaconazole oral suspension 18 mg/kg/day divided into 3 doses (TID) until recovery from neutropenia or up to 28 days.
- POS 18 TID 7 to <18 Yrs: Participants aged 7 to <18 years received posaconazole oral suspension 18 mg/kg/day divided into 3 doses (TID) until recovery from neutropenia or up to 28 days.
- POS 12 TID 3 Months to <2 Yrs: Participants aged 3 months to <2 years received posaconazole oral suspension 12 mg/kg/day divided into 3 doses (TID) until recovery from neutropenia or up to 28 days.
Arm/Group | POS 12 BID 2 to <7 Yrs | POS 12 BID 7 to <18 Yrs | POS 18 BID 2 to <7 Yrs | POS 18 BID 7 to <18 Yrs | POS 18 TID 2 to <7 Yrs | POS 18 TID 7 to <18 Yrs | POS 12 TID 3 Months to <2 Yrs
Serious Adverse Events (participants affected / at risk) | 5/22 | 3/21 | 1/19 | 7/28 | 7/15 | 11/30 | 1/1
Other Adverse Events (participants affected / at risk) | 21/22 | 20/21 | 16/19 | 26/28 | 13/15 | 28/30 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | POS 12 BID 2 to <7 Yrs (N=22) | POS 12 BID 7 to <18 Yrs (N=21) | POS 18 BID 2 to <7 Yrs (N=19) | POS 18 BID 7 to <18 Yrs (N=28) | POS 18 TID 2 to <7 Yrs (N=15) | POS 18 TID 7 to <18 Yrs (N=30) | POS 12 TID 3 Months to <2 Yrs (N=1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 5 (7) | 5 (5) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic haemorrhage (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic vein occlusion (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary disease (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venoocclusive liver disease (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Puncture site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chemotherapeutic drug level increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burkitt's lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | POS 12 BID 2 to <7 Yrs (N=22) | POS 12 BID 7 to <18 Yrs (N=21) | POS 18 BID 2 to <7 Yrs (N=19) | POS 18 BID 7 to <18 Yrs (N=28) | POS 18 TID 2 to <7 Yrs (N=15) | POS 18 TID 7 to <18 Yrs (N=30) | POS 12 TID 3 Months to <2 Yrs (N=1)
Anaemia (Blood and lymphatic system disorders) | 4 (6) | 2 (3) | 3 (6) | 8 (12) | 3 (11) | 6 (12) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 4 (4) | 0 (0) | 4 (4) | 4 (5) | 5 (5) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3/4 (3) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (19) | 7 (15) | 3 (10) | 6 (22) | 1 (2) | 5 (8) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 3 (4) | 0 (0)
Antithrombin III deficiency (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Eye movement disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 6 (7) | 1 (1) | 2 (2) | 3 (3) | 4 (5) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 4 (5) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 3 (3) | 3 (5) | 7 (7) | 3 (7) | 5 (5) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Loose tooth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (8) | 3 (3) | 2 (5) | 9 (9) | 3 (3) | 13 (21) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 3 (4) | 0 (0) | 2 (2) | 4 (5) | 5 (9) | 6 (8) | 0 (0)
Tongue coated (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 8 (13) | 3 (5) | 5 (6) | 11 (14) | 7 (11) | 9 (14) | 0 (0)
Catheter site erythema (General disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Catheter site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Device occlusion (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 6 (7) | 0 (0)
Mucosal inflammation (General disorders) | 9 (9) | 3 (3) | 2 (5) | 7 (7) | 1 (1) | 4 (4) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 13 (14) | 8 (9) | 3 (3) | 8 (10) | 2 (4) | 6 (7) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Engraftment syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Graft versus host disease in skin (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alpha haemolytic streptococcal infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pseudomonal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Procedural headache (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 2 (5) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (5) | 1 (1) | 0 (0)
Biopsy skin (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (3) | 0 (0)
Fluid balance positive (Investigations) | 1 (1) | 3 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (3) | 2 (4) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 2 (11) | 1 (1) | 2 (5) | 4 (11) | 0 (0)
Transaminases increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (3) | 3 (4) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 8 (9) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hyperalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 3 (3) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (6) | 1 (1) | 1 (2) | 4 (6) | 2 (3) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (2) | 0 (0) | 2 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (4) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 8 (10) | 1 (1) | 3 (3) | 0 (0)
Abnormal behavior (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Genital rash (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus genital (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 3 (3) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 3 (4) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5) | 1 (1) | 3 (5) | 2 (5) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 2 (3) | 4 (5) | 2 (2) | 5 (5) | 0 (0)
Red man syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Central venous catheter removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Central venous catheterisation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 4 (5) | 1 (1) | 1 (1) | 3 (3) | 2 (3) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 0 (0)
Venoocclusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Local swelling (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital ulceration (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Penile oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Only 1 participant was enrolled in the POS 12 TID 3 months to <2 years group, limiting conclusions that may be drawn for pharmacokinetics or safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the study. The sponsor shall have the right to review and comment with respect to publications, abstracts, slides, and manuscripts and the right to review and comment on the data analysis and presentation with regard to proprietary information, accuracy, fair balance, and compliance.